CLINICAL TRIAL: NCT04360915
Title: Assessing the Pharmacokinetics Effects of Food on ASK120067 in Single Oral Administration in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASK-LC-120067-Ib
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASK120067 in fast condition (Experimental): Take ASK120067 tablets orally once in the first day at 160mg in fast condition.
  Interventions: Drug: ASK120067
- ASK120067 in fed condition (Experimental): Take ASK120067 tablets orally once in the first day at 160mg in fed condition.
  Interventions: Dietary Supplement: ASK120067 in fed condition

INTERVENTIONS:
Drug: ASK120067 — Take ASK120067 tablets orally in first day at 160 mg in fast condition.
  Arms: ASK120067 in fast condition
Dietary Supplement: ASK120067 in fed condition — Take ASK120067 tablets orally in first day at 160 mg in fed condition.
  Arms: ASK120067 in fed condition

SUMMARY:
To evaluate the pharmacokinetic characteristics of ASK120067 and CCB4580030 after the single oral administration of ASK120067 in fast and after a high-fat meal in healthy Chinese subjects, and to evaluate the effect of food on the bioavailability of ASK120067.To evaluate the safety of ASK120067 tablets administered orally in fast and fed.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy subjects aged 18 or above and 45 or below, male and female;
* 2) The weight of male subjects shall not be less than 50 kg, and that of female subjects shall not be less than 45 kg.Body mass index (BMI) = weight (kg)/height2 (m2), BMI = Within the range of 19.0~26.0 (including the critical value);
* 3) Normal or abnormal physical examination (physical examination, vital signs, laboratory examination, 12-lead electrocardiogram, frontal and lateral chest radiographs, etc.) during the screening period has no clinical significance;
* 4) Subjects (including male subjects) are willing to have no pregnancy plan from the screening date to 6 months after the last dose, and are willing to take effective contraceptive measures;
* 5) Subjects should sign the informed consent before the test, fully understand the test content, process and possible adverse reactions, have good communication with researchers and complete the test according to the test plan.

Exclusion Criteria:

* 1) patients with clinical significance who are abnormal by comprehensive physical examination, vital signs examination, routine laboratory examination (blood routine, urine routine, blood biochemistry, coagulation function), 12-lead electrocardiogram, and positive and lateral chest radiographs;
* 2) HBSAg HCVAb HIVAb, treponema palliatum antibody and other test results were positive;
* 3) QTc interphase abnormality (QTc>450ms) with clinical significance;
* 4) participated in the drug clinical trial within 3 months before the trial;
* 5) taking any medication 14 days before the trial;
* 6) surgical resection history, such as: hepatectomy, nephrectomy, digestive organ (gallbladder) resection;
* 7) history of tuberculosis;
* 8) past history of deep vein thrombosis/other thromboembolic events, abnormal coagulation factors, thrombocytopenia, or abnormal platelet function;
* 9) previous history of interstitial lung disease (ILD), drug-induced ILD, radioactive pneumonia requiring steroid treatment, or clinically active ILD with evidence;
* 10) allergic or hypersensitive to ASK120067 experimental active ingredients or inactive excipients, drugs with similar chemical structure to the experimental drugs or drugs with the same target, allergic to two or more drugs and food;
* 11) there are swallowing difficulties or gastrointestinal diseases affecting drug absorption;
* 12) have any disease that increases the risk of bleeding, such as acute gastritis or gastric and duodenal ulcers;
* 13) habitual constipation or diarrhea;
* 14) heavy drinking and/or a history of excessive drinking (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
* 15) alcohol breath test > 0.0mg /100mL;
* 16) drug abuse screening positive;
* 17) smoking history, smoking more than 5 cigarettes per day in the first 3 months of the screening period or habitual use of nicotine-containing products, and unable to quit during the trial;
* 18) those with positive urine nicotine detection results at the screening stage;
* 19) having a history of blood or needle sickness;
* 20) habitual consumption and consumption of special diet (including grapefruit juice, star fruit, pitaya fruit, etc.) within 7 days before the test, or the presence of other factors affecting drug absorption, distribution, metabolism, excretion, etc.;
* 21) blood donation or massive blood loss (> 400 mL) within 3 months prior to the trial;
* 22) an acute illness or accident occurs during the screening period;
* 23) the female subjects were lactating, or the pregnancy test results were positive, or they had unprotected sex within 2 weeks before the screening date;
* 24) there are other conditions that the researcher thinks are not suitable for inclusion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples will be collected from each subject at pre-specified times after the administration of the study on Day 1, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out maximum concentration
AUC | Blood samples will be collected from each subject at pre-specified times after the administration of the study on Day 1, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out area under the plasma concentration-time curve

SECONDARY OUTCOMES:
Tmax | Blood samples will be collected from each subject at pre-specified times after the administration of the study on Day 1, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out time to reach maximum concentration
t1/2 | Blood samples will be collected from each subject at pre-specified times after the administration of the study on Day 1, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out apparent end elimination half-life
CL/F | Blood samples will be collected from each subject at pre-specified times after the administration of the study on Day 1, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out apparent clearance
Vd/F | Blood samples will be collected from each subject at pre-specified times after the administration of the study on Day 1, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out apparent volume of distribution
λz | Blood samples will be collected from each subject at pre-specified times after the administration of the study on Day 1, (pre-dose, 0.25h,0.5h, 1h,1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 5h, 6h, 8h, 12h, 24h,36h,48h,72 hours post dose)
  Collect plasma concentrations of ASK120067 and 1 metabolites following single dose at designated time points of Day 1 to figure out apparent terminal elimination rate constant
Incidence and Severity of Treatment-Emergent Adverse Events | Adverse events will be collected from baseline until 12 days after the administration and the follow-up period
  Assessed by number and severity of adverse events as recorded on the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Zourong Ruan, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided